CLINICAL TRIAL: NCT04068363
Title: Donor Gender Effect on Graft Function in Adult Egyptian Patients Undergoing Living Donor Liver Transplant: A Single Centre Retrospective Study
Brief Title: Donor Gender Effect on Graft Function in Adult Egyptian Patients Undergoing Living Donor Liver Transplant
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: IBR/0006379
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Donor to Recipient Gender Mismatch in LDLT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Matched group: Same sex of both donor and recipient
  Interventions: Other: non interventional
- Mismatched group: Sex mismatch between donor and recipient, subgroups might be added
  Interventions: Other: non interventional

INTERVENTIONS:
Other: non interventional — non interventional study

SUMMARY:
Liver transplantation (LT) represents the gold-standard therapy for the treatment in case of dreadful liver pathologies . It is thus a main concern to optimize the results in terms of post-LT survivals. The effect of gender match on post-transplant outcome is still debatable. Hormonal , and size difference between female and male may be proposed to affect the post transplant outcome . The aim of this study is to evaluate the effect of donor-recipient gender mismatch on survival rates

ELIGIBILITY:
Inclusion Criteria:

* Adult Egyptian Patients >18 years.

Exclusion Criteria:

* Patient refusal.
* Patients who underwent re-transplantation before discharge from the ICU after the first liver transplant.
* Intraoperative cardiac arrest or immediately postoperative cardiac arrest within the first 6 hours postoperative.
* Massive blood loss.
* Pre-existing renal failure requiring hemodialysis or continuous hemofiltration.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intraoperatively, Both standard anesthetic and piggyback liver transplant for hepatic transplantation will be performed by the same anesthesia and surgical team . Intraoperative hemodynamics (MAP and HR), graft weight to recipient weight ratio (GWRWR), blood products transfused and intraoperative adverse events will be recorded. At the end of surgery patients will be transferred to the ICU where they will be monitored and will receive the standard protocol for postoperative management after liver transplantation.
  - Recipients will be divided into two groups ( matched and mismatched) and will be subdivided based on the following variables: recipient age, MELD score, intraoperative packed red blood cells (PRBC) and fresh frozen plasma (FFP) transfusions, duration of cold ischemia. These subgroups will be compared with respect to 2-year graft survival separately in recipients of sex matched and mismatched transplantation.
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
2 years survival post liver transplant. | 3 months
  The primary outcome will be survival at 2 years post liver transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No